CLINICAL TRIAL: NCT06887790
Title: An Investigation of the Effect of the Ethics Course Based on the Arcs Model on Achievement, Academic Self-efficacy and the Effectiveness of Education in Ethics
Brief Title: Success, Academic Self-efficacy; ARCS Model
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Güzel Nur Yıldız, Dr, Assoc. Prof., Muş Alparslan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: MusAlparslanU
Record Dates: First submitted 2025-02-22; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Success Rate; Self-Efficacy
Keywords: Success, self-efficacy, ethics training, ARCS
MeSH Terms: conditions — Arthrogryposis renal dysfunction cholestasis syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARCS Group (Experimental): The experimental group will be given structured training with the ARCS method.
  Interventions: Other: Education method (ARCS)
- Control Group (No Intervention): The control group will not be intervened in the study.

INTERVENTIONS:
Other: Education method (ARCS) — The control group will not be intervened in the study. The experimental group will be given structured training with the ARCS method.
  Arms: ARCS Group

SUMMARY:
Cassels and Redman have offered some suggestions such as teaching students basic ethical principles and theories, the International Council of Nurses (ICN) Code of Ethics, and the rights and laws of nurses in all kinds of ethical issues they may encounter in practice in order to increase their ethical decision-making skills. When the academic literature is examined, it is seen that ethics education has positive effects on the development of nursing students. Ethics education in nursing from a multi-dimensional perspective is very important in determining the quality of education and restructuring education. According to Bandura, self-efficacy is based on our belief in our abilities and is necessary to organize and demonstrate a behavior necessary to achieve our goals. In today's world where the quality and structure of education are seriously discussed, the importance of these evaluations in terms of university education is rapidly increasing. When researching the increase in quality in education, it is important to consider the individual's perspective on his/her own abilities as well as social abilities and to accept this as an important element of the individual's ability to act. Self-efficacy, which is one of the concepts that comes to the fore when the individual's self-predictions and evaluations are expressed, should also be addressed in relation to university education.

DETAILED DESCRIPTION:
Ethical decision-making requires knowledge and management skills about ethical theories, ethical principles and practices. Therefore, ethics education for nurses is extremely important, especially at undergraduate and graduate levels, in practical professional life. Otherwise, only an intuitive path will be followed in the ethical decision-making process and professionalism will be abandoned. In recent years, ethics education has gained great importance in nursing education and more contemporary models (such as clinical practice models, case studies) have begun to be integrated in education so that nurses can participate in the ethical decision-making process. Cassels and Redman have offered some suggestions for students to increase their ethical decision-making skills, such as teaching them basic ethical principles and theories, the International Council of Nurses (ICN) Code of Ethics, and the rights and laws of nurses in all kinds of ethical problems they may encounter in practice. When the academic literature is examined, it is seen that ethics education has positive effects on the development of nursing students. In addition, nursing students also state that ethics education is an important part of their undergraduate education. On the other hand, studies have shown that nurses do not feel prepared to solve ethical problems in practice. This raises the question of whether ethics education in nursing is sufficiently effective in developing ethical knowledge and skills of nursing students in terms of method and content. Because, effective measurement, evaluation and feedback of learning outcomes and behavioral changes in students are important factors in the learning process. When the literature is examined; various surveys have been used to examine the effectiveness of ethics education in nursing students. Some of these focused on the theoretical content of ethics education, while others focused on specific methods used in education. In some surveys, only the satisfaction levels of students with ethics education were determined. However, evaluating the effectiveness of ethics education in nursing from multiple perspectives is very important in determining the quality of education and restructuring education. In this way, nursing students who receive qualified ethics education can develop a certain ethical awareness and sensitivity, and they can be provided with responsibility in ethical decision-making. The concept of self-efficacy is frequently applied, especially in processes related to education - for example, in terms of learning and performance - to combat stress and investigate the physical health status of teachers and students. Self-efficacy expectation is defined as "the person's self-convincing about their abilities". It is reported that positive self-efficacy expectations increase motivation, enable the person to cope with new and difficult tasks, and make them willing to make an effort; whereas negative self-efficacy expectations cause the person to fail to act on their own initiative or to leave a task unfinished. Self-efficacy belief is defined as "the belief that an individual has in their capacity to organize and successfully perform the necessary activity to demonstrate a certain performance". According to Bandura, self-efficacy is based on our belief in our abilities and is necessary to organize and demonstrate a behavior necessary to achieve our goals. In today's world where the quality and structure of education are seriously discussed, the importance of these evaluations in terms of university education is rapidly increasing. While researching the increase in quality in education, the view that the individual's perspective on their own abilities should be taken into consideration in addition to social abilities and that this should be accepted as an important element of the individual's ability to act is gaining importance. Self-efficacy, which is one of the prominent concepts when the individual's self-predictions and evaluations are expressed, should also be addressed in relation to university education.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Being educated in the nursing program,
* Not having taken the "Nursing Ethics" course before,
* Not being absent during the data collection processes.
* Having a phone and internet connection that can enter Google forms.

Exclusion Criteria:

* Being absent during the research process,
* Dropping from education,
* Not cooperating, Protocol registration

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-04-02 (Estimated)

PRIMARY OUTCOMES:
achievement test | 1 month
  achievement test average

CONTACTS AND LOCATIONS:
Overall Officials: Guzel Nur YILDIZ, Associate Proof., Principal Investigator — Mus Alparslan Univercity
Locations (1):
- Muş Alparslan University, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In order to determine the privacy of individuals.